CLINICAL TRIAL: NCT06768749
Title: The Impact of Melatonin Lotion on Actigraphy, Sleep Quality, Autonomic Nervous System Indicators, Mood, Anxiety Symptoms, and Side Effects
Brief Title: The Impact of Melatonin Lotion on Sleep and Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Redlands (Other)
Responsible Party: Principal Investigator, Lisa Olson, Professor of Biology, University of Redlands
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024-032
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Sleep Problems; Depressive Disorder and Anxiety Disorders
Keywords: melatonin; sleep; heart rate variability; actigraphy; amylase; mood; anxiety; depression
MeSH Terms: conditions — Parasomnias; Depressive Disorder; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin lotion first (Experimental): Participants will be randomized to one week of treatment with melatonin lotion, followed by a week washout, then one week of treatment with placebo lotion
  Interventions: Other: Melatonin lotion; Other: Placebo lotion
- Placebo lotion first (Experimental): Participants will be randomized to one week of treatment with placebo lotion, followed by a week washout, then one week of treatment with melatonin lotion
  Interventions: Other: Melatonin lotion; Other: Placebo lotion

INTERVENTIONS:
Other: Melatonin lotion — 3 g lotion applied one hour before bedtime
Other: Placebo lotion — 3 g of placebo lotion (scent-matched control) applied one hour before bedtime

SUMMARY:
The purpose of this study is to examine the effect that melatonin lotion has on sleep quality, the nervous system, and mental health. Melatonin is a hormone secreted by the brain that regulates sleep and might improve depression and anxiety symptoms. The goal is to determine whether melatonin in lotion form is an effective treatment for young adults with inadequate sleep and might improve mental health. Participants will fill out surveys, wear an actigraph (a wrist-worn device that measures sleep), wear a heart rate monitor (a strap worn around one's chest), and provide nightly saliva samples during treatment weeks. In one of the two treatment weeks, participants will receive a lotion that contains melatonin. During the other week they will receive a control treatment that will be lotion with no melatonin, and there will be a week in between with no treatment at all.

DETAILED DESCRIPTION:
All participants will receive a melatonin lotion and a placebo lotion in a randomized crossover design. Participants will receive equipment and supplies on a Monday and will begin the assigned treatment that night, by self-applying premeasured lotion 1 hour before bedtime. During the two treatment weeks, participants will wear ActiGraph GT3X-BT accelerometers (ActiGraph, Pensacola, FL) at all times except when bathing or submerged in water. They will wear Polar H10 heart rate monitor chest straps (Polar Electro, Kempele, Finland) from one hour prior to bedtime until after a 5 min sitting period after waking. Three times daily they will be asked 1-item mood/anxiety questions ("How ___ do you feel right now?") through REDCap software. Participants will check any experienced side effects off a checklist once daily. Participants will collect a passive drool sample daily at bedtime and store in their home freezer until returning the samples to the laboratory. Treatment will occur for seven nights, with a return of equipment and saliva samples as well as confirmation of actigraphy and HRV readings the following Monday. After a seven day washout period to reduce any carryover effects, equipment and supplies will be supplied the next Monday and the participant will begin the other assigned treatment (active or placebo) that night in a crossover design. At three timepoints (pre-treatment, at the end of the melatonin treatment week, and at the end of the placebo week), participants will answer the following surveys online via REDCap: PROMIS short forms for anxiety, depression, sleep quality, and sleep-related impairment.

ELIGIBILITY:
Inclusion Criteria:

* a T score ≥ 48 on the sleep disturbance short form Patient-Reported Outcomes Measurement Information System (PROMIS) measure, and
* a T score ≥ 55 on the anxiety or depression short form PROMIS measures (mild symptoms or more)

Exclusion Criteria:

* currently using antidepressant, anti-anxiety, or sleep medication including melatonin
* are pregnant
* have allergies/sensitivities to scented lotion
* are unwilling to commit to keeping a similar bedtime (± 1 hour) during treatment weeks.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Sleep disturbance | Measured pre-treatment, at end of placebo week, and at end of active treatment week (3 weeks total)
  PROMIS SF v1.0 - Sleep Disturb 8b
Anxiety | Measured pre-treatment, at end of placebo week, and at end of active treatment week (3 weeks total)
  PROMIS SF v1.0 - Anxiety 8a
Depression | Measured pre-treatment, at end of placebo week, and at end of active treatment week (3 weeks total)
  PROMIS SF v1.0 - Depression 8b
Total sleep time | Two weeks of data separated by a one week period
  Measured via actigraphy
Sleep efficiency | Two weeks of data separated by a one week period
  Measured by actigraphy
Normalized high frequency power of heart rate variability | Two weeks of data separated by a one week period
  5 min period during sleep latency, overnight recording while sleeping, and 5 min period sitting upright each morning
Anxiety by momentary ecological assessment | Three times per day for two weeks of data separated by a one week period
  One item question: "How anxious do you feel right now?"
Mood by momentary ecological assessment | Three times per day for two weeks of data separated by a one week period
  Single-item questions ("How ___ do you feel right now?)
Salivary alpha-amylase | Daily at bedtime for two weeks of data separated by a one week period
  As an indicator of sympathetic nervous system activity

SECONDARY OUTCOMES:
Sleep-related impairment | Measured pre-treatment, at end of placebo week, and at end of active treatment week (3 weeks total)
  PROMIS SF v1.0 - Sleep-Related Impairment 8a
Other sleep variables | Two weeks of data separated by a one week period
  A MANOVA will be conducted with the primary sleep outcomes as well as sleep onset latency (both self-reported and as measured by actigraphy) and subjective sleep quality
Salivary melatonin | Daily at bedtime for two weeks of data separated by a one week period
  For confirmation of protocol compliance
Other HRV variables | 5 min period sitting upright each morning after waking, and overnight data capture starting one hour before bedtime
  A MANOVA will be conducted with autonomic nervous system indicators including normalized high frequency HRV and salivary alpha amylase as primary outcomes, but also including LF/HF ratio, RMSSD, and pNN50
Side effects | Daily for two weeks of data separated by a one week period
  Frequency of headache, drowsiness, skin irritation, vivid dreams, nightmares, dizziness, and other

CONTACTS AND LOCATIONS:
Overall Officials: Lisa E Olson, Ph.D., Principal Investigator — University of Redlands
Locations (1):
- University of Redlands, Redlands, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD (deidentified through the safe harbor method)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be submitted after publication of the main study outcomes, and will remain on the National Sleep Research Resource server indefinitely
Access Criteria: Data will be provided via the National Sleep Research Resource and access allowed according to their criteria